CLINICAL TRIAL: NCT06571565
Title: Manual Lymph Drainage in Fibromyalgia Patients; Oxidative Stress, Pain, Functional Effect on Mood and Sleep Quality
Brief Title: The Effect of Manual Lymph Drainage in Fibromyalgia Patients
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PDANALAN
Record Dates: First submitted 2024-08-05; First posted 2024-08-26 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-08

CONDITIONS: Fibromyalgia; Oxidative Stress
Keywords: Fibromyalgia; manual lymph drainage; lymph; oxidative stress
MeSH Terms: conditions — Fibromyalgia | interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: As a randomized controlled single blind
Who Masked: Investigator
Masking Description: The evaluator and the researcher working on the antioxidant panel will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- working group (Experimental): Conservative treatment will be applied to the back-neck region. In this treatment, 20 min hotpack, 10 min ultrasound agent (frequency 0.5-3.5MHz), 20 min Transcutaneous Electrical Nerve Stimulation (TENS) agent (Conventional TENS; Frequency 60-80 Hz, current passage time 50-100 microseconds) will be given. 15 sessions will be applied. Unlike the control group, manual lymph drainage treatment, the effect of which is aimed to be investigated, will be applied to the study group. Manual lymph drainage treatment will be performed by a lymphedema physiotherapist trained in Manual Lymph Drainage / Complex Unloading Physiotherapy.
  Interventions: Combination Product: conservative treatment
- control group (Active Comparator): Conservative treatment will be applied to the back-neck region. In this treatment, 20 min hotpack, 10 min ultrasound agent (frequency 0.5-3.5MHz), 20 min Transcutaneous Electrical Nerve Stimulation (TENS) agent (Conventional TENS; Frequency 60-80 Hz, current passage time 50-100 microseconds) will be given. 15 sessions will be applied.
  Interventions: Combination Product: conservative treatment

INTERVENTIONS:
Combination Product: conservative treatment — Conservative treatment will be applied to the back-neck region in both groups. In this treatment, 20 min hotpack, 10 min ultrasound agent (frequency 0.5-3.5MHz), 20 min Transcutaneous Electrical Nerve Stimulation (TENS) agent (Conventional TENS; Frequency 60-80 Hz, current passage time 50-100 microseconds) will be given.

SUMMARY:
In this randomized controlled single blinded study, our primary objective is to evaluate the effects of manual lymphatic drainage on blood lipid peroxidation system and antioxidant system in FMS patients. For this objective, the following biochemical analyses will be performed to objectively evaluate the effect of manual lymphatic drainage.

Our secondary objective is to evaluate the changes in pain, functional status and sleep quality with manual lymphatic drainage treatment. The evaluator and the investigator working on the antioxidant panel will be blinded.

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) is a chronic musculoskeletal disorder with poorly understood pathophysiology and etiology, characterized by tender points in specific anatomical regions, often accompanied by fatigue, cognitive impairment, psychiatric symptoms, sleep disturbances and multiple somatic symptoms. FMS is a difficult disease to treat and may require the use of multifaceted treatment modalities. The main goal of treatment is to reduce pain, regulate sleep and improve physical function. There are different results in studies investigating the effectiveness of treatment modalities in FMS and there is no standardization in the methodology of these studies. In randomized controlled trials and systematic reviews, there is moderate evidence that massage improves sleep quality and reduces anxiety. In the literature, lymph drainage has been applied to these patients as a treatment method and there is limited evidence that it reduces pain.

In this randomized controlled single blinded study, our primary objective was to evaluate the effects of manual lymphatic drainage on blood lipid peroxidation system and antioxidant system in FMS patients. For this objective, the following biochemical analyses will be performed to objectively evaluate the effect of manual lymphatic drainage.

Our secondary objective is to evaluate the changes in pain, functional status and sleep quality with manual lymphatic drainage treatment. The evaluator and the researcher working on the antioxidant panel will be blinded. The study will include female patients aged 25 years and older, who have been diagnosed with FMS for at least 2 years and whose level of medication use for FMS treatment has been stable for at least 3 months, who apply to Başkent University Adana Research and Application Center Physical Therapy and Rehabilitation clinic for fibromyalgia syndrome treatment.

Patients will be evaluated in terms of pain intensity, sleep, functional status and quality of life as well as oxidative stress and antioxidant levels in three stages: before treatment, immediately after treatment and one month after the end of treatment. Blood samples will be taken before treatment, immediately after treatment and one month after treatment for the evaluation of oxidative stress and antioxidant levels. Paraoxonase (PON1), Oxidative Stress Index (OSI), Malondialdehyde (MDA), Reduced Glutathione (GSH), Low Density Lipoprotein (LDL), High Density Lipoprotein (HDL) and Triglyceride levels will be analyzed in these blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 25 years and older who have been admitted to the Physical Therapy and Rehabilitation clinic for the treatment of fibromyalgia syndrome, who have been diagnosed with FMS for at least 2 years and whose medication use level for FMS treatment has been stable for at least 3 months will be included.

Exclusion Criteria:

* The exclusion criteria were determined as follows: Patients with concomitant decompensated and/or acute cardiovascular disease, scar tissue that disrupts the integrity of the skin in the area of application (back-neck), use of psychiatric medication (recently started or ongoing psychiatric medical treatment for less than 3 months, antipsychotic treatment that has not yet reached the therapeutic dose), acute infection of bacterial or viral origin.

In addition, people with uncontrolled additional rheumatologic diseases that may affect the patient's pain, sleep, functional status and anti-oxidant biochemical parameters, and people with endocrinometabolic diseases such as hypothyroidism, which may change the soft tissue structure in the treatment area and cause edema, will be excluded from the study.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 25 years and older
Enrollment: 44 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
oxidative stress and other biochemical analyzes | Both groups will be evaluated before treatment, immediately after treatment and one month after treatment.
  To evaluate the effects of manual lymphatic drainage on blood lipid peroxidation system and antioxidant system in FMS patients. For this objective, the following biochemical analyses will be performed to objectively evaluate the effect of manual lymphatic drainage.Blood samples will be taken from the patients before, after and one month after the end of treatment and Paraoxonase (PON1), Oxidative Stress Index (OSI), malondialdehyde (MDA), Rductegulutathione (GSH), Low danditelilipoprotein (LDL), High danditelilipoprotein (HDL) and Triglyceride levels will be evaluated.

SECONDARY OUTCOMES:
Pain evaluation of | Both groups will be evaluated before treatment, immediately after treatment and one month after treatment.
  Pain will be assessed with the Mcgill-Melzack pain questionnaire.
Functional Status evaluation of | Both groups will be evaluated before treatment, immediately after treatment and one month after treatment.
  Quality of life and functional status will be assessed with the Fibromyalgia Impact Questionnaire (FEA).
Sleep quality evaluation of | Both groups will be evaluated before treatment, immediately after treatment and one month after treatment.
  Sleep quality will be assessed with the Pittsburgh Sleep Inventory (PSI). The PDQI is a scale that provides information about sleep quality and the type and severity of sleep disturbance in the last month.

CONTACTS AND LOCATIONS:
Overall Officials: Selen OZGOZEN, Dr, Study Chair — dr
Locations (1):
- Baskent University, Adana, çukurova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The evaluator and the researcher working on the antioxidant panel will be blinded.

REFERENCES:
- [Background] Bennett RM, Friend R, Marcus D, Bernstein C, Han BK, Yachoui R, Deodhar A, Kaell A, Bonafede P, Chino A, Jones KD. Criteria for the diagnosis of fibromyalgia: validation of the modified 2010 preliminary American College of Rheumatology criteria and the development of alternative criteria. Arthritis Care Res (Hoboken). 2014 Sep;66(9):1364-73. doi: 10.1002/acr.22301. PMID 24497443
- [Background] Heidari F, Afshari M, Moosazadeh M. Prevalence of fibromyalgia in general population and patients, a systematic review and meta-analysis. Rheumatol Int. 2017 Sep;37(9):1527-1539. doi: 10.1007/s00296-017-3725-2. Epub 2017 Apr 26. PMID 28447207